CLINICAL TRIAL: NCT06041880
Title: To Stretch, Not Strain: Impact of Passive Stretching on Calf Muscle and Gait Mechanics in PAD
Brief Title: Passive Calf Stretching Therapy in Peripheral Artery Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, David N. Proctor, PhD, Principal Investigator, Penn State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 00022960
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Artery Disease; Claudication, Intermittent
Keywords: Endothelial dysfunction
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to 4-weeks of stretching or no stretching. Following the first 4-week intervention, participants will crossover and perform whichever intervention they did not receive previously.
Masking Description: Due to the nature of the intervention, participants will not be blinded to stretching vs no-stretching interventions. The study team will be blinded to intervention order when performing data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- 4-weeks of passive calf stretching for 30 minutes 5 days a week (Experimental): A modified plantar fasciitis ankle splint will be used to passively stretch the calf muscle.
  Interventions: Device: Passive calf muscle stretching device
- 4-weeks of no-stretching (No Intervention): No device will be used to stretch the calf muscle. Participants will go about their normal daily activity for 4-weeks.

INTERVENTIONS:
Device: Passive calf muscle stretching device — Modified night splints will be used to passive stretch the calf muscle.
  Other Names: Plantar fasciitis night splints
  Arms: 4-weeks of passive calf stretching for 30 minutes 5 days a week

SUMMARY:
The goal of this clinical trial is to assess the effects of passive calf muscle stretching in patients diagnosed with peripheral artery disease (PAD). The main question it aims to answer are:

1. To determine if daily calf muscle stretching at home improves calf muscle and vascular health.
2. To determine if daily calf muscle stretching at home improves walking performance.

Participants will use inflatable ankle splints for 30 minutes a day, 5 days a week for 4-weeks on both days and 4-weeks of no stretching.

DETAILED DESCRIPTION:
Patients with peripheral artery disease will passively stretch their calf muscles using a stretch device on both feet for 30 minutes a day for 4 weeks. Blood vessel health and size, length and function of the calf muscles and tendons and walking performance will be measured. Joint and foot movements as well as calf muscle oxygen levels will be measured during walking performance tests.

ELIGIBILITY:
Inclusion Criteria:

* Presence of PAD
* Stable condition (PAD symptoms) for at least 3 months
* Age 40-85
* Men and women who are not pregnant or nursing

Exclusion Criteria:

* Ischemic leg pain at rest; critical limb ischemia (ulceration or gangrene)
* Any condition other than PAD that limits the ability to walk
* Major surgery or lower extremity revascularization surgery in the past 6 months
* Myocardial infarction within past 6 months or unstable angina
* Severe lung disease (on supplemental oxygen or frequently use rescue inhalers)
* Participants with non-compressible vessels (ABI > 1.40)
* Habitual exercise (30 minutes of continuous activity on 3 or more days per week)
* Current tobacco smoker or use of nicotine-containing products
* Pregnant or nursing women
* History or ankle reconstruction or surgery Recent history (<1 year) of injuries to the ankle, Achilles tendon, or feet
* History of rheumatoid arthritis or other degenerative joint disease
* Major medical illness treatment during the prior 12 months
* Uncontrolled hypertension
* Uncontrolled diabetes
* Inability to walk on a treadmill at a slow pace (1.0 mile/hour)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test distance | 6-12 minutes
  Submaximal exercise test used to assess aerobic capacity and endurance
Muscle to tendon ratio | 45 minutes
  The ratio of gastrocnemius muscle fascicle length to Achilles' tendon length will be measured using ultrasound
Endothelial function | 30 minutes
  Popliteal flow-mediated dilation will be measured as a index of macrovascular endothelial function in the leg.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No